CLINICAL TRIAL: NCT05737511
Title: Efficacy of Hydroxyzine Versus Treatment as Usual for Panic Disorder: An Eight-Week, Open Label, Pilot, Randomized Controlled Trial.
Brief Title: Efficacy of Hydroxyzine for Patients With Panic Disorder
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sultan Qaboos University (Other)
Responsible Party: Principal Investigator, Mohammed Al Alawi, Principal Investigator, Dr Mohmmed Al Alawi Bsc, MD,PhD, MRCPsych, OMSBPsych, ARABPsych, Sultan Qaboos University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 02/2023
Record Dates: First submitted 2023-02-10; First posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Panic Disorder
MeSH Terms: conditions — Panic Disorder | interventions — Hydroxyzine; Escitalopram; Citalopram; Fluoxetine; Fluvoxamine; Paroxetine; Sertraline; Alprazolam; Clomipramine; Clonazepam; Diazepam; Imipramine; Lorazepam; Mirtazapine; Reboxetine; Valproic Acid; Duloxetine Hydrochloride; Gabapentin; Levetiracetam; Milnacipran; Moclobemide; Olanzapine; Phenelzine; Quetiapine Fumarate; Risperidone; Tranylcypromine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydroxyzine (Experimental): Hydroxyzine (25 mg/day) for eight weeks, the dose of hydroxyzine may be adjusted based on tolerability and clinical judgment, max 100mg/day
  Interventions: Drug: Hydroxyzine
- Treatment as Usual (Active Comparator): Treatment as usual includes the currently approved treatment according to CANMAT and Muadesly guidelines
  Interventions: Drug: Escitalopram Oxalate

INTERVENTIONS:
Drug: Hydroxyzine — Oral tablet of hydroxyzine 25mg at night which could be increased to TID or QID
  Other Names: Atarax; Vistaril
  Arms: Hydroxyzine
Drug: Escitalopram Oxalate — The treatment as usual can include first-line, second-line and third-line recommendations
  Other Names: citalopram; fluoxetine, fluvoxamine, paroxetine, paroxetine CR, sertraline, venlafaxine XR,; Alprazolam, clomipramine, clonazepam, diazepam, imipramine, lorazepam, mirtazapine, reboxetine; Bupropion SR, divalproex, duloxetine, gabapentin, levetiracetam, milnacipran, moclobemide, olanzapine, phenelzine, quetiapine, risperidone, tranylcypromine
  Arms: Treatment as Usual

SUMMARY:
The aim of this study is to evaluate the efficacy of hydroxyzine compared to treatment as usual (TAU) for patients with panic disorder. By conducting a pilot study, we hope to provide initial data on the feasibility and potential impact of hydroxyzine for this population. This will inform the design and power calculations of a larger, more comprehensive study in the future.

Objectives:

To assess the feasibility of conducting a randomized controlled trial (RCT) of hydroxyzine for panic disorder.

To evaluate the effectiveness of hydroxyzine compared to TAU in reducing panic symptoms in patients with panic disorder.

To explore the potential side effects and tolerability of hydroxyzine in this population.

Methods:

This will be a single-center, open-label, randomized pilot study. A total of 30 patients with a primary diagnosis of panic disorder will be recruited from a psychiatric outpatient clinic. Participants will be randomly assigned to receive either hydroxyzine or TAU for 8 weeks. The primary outcome measure will be the change in panic symptoms as assessed by the Panic Disorder Severity Scale (PDSS). Secondary outcome measures will include the Hamilton Anxiety Rating Scale (HAM-A) and the Clinical Global Impression-Severity (CGI-S) scale. Participants will be assessed at baseline, 4 weeks, and 8 weeks. Adverse events will be monitored throughout the study.

Expected Results:

This pilot study is expected to provide preliminary data on the feasibility and potential efficacy of hydroxyzine for panic disorder. The results will inform the design of a larger RCT to further evaluate the efficacy of hydroxyzine for this population.

Significance:

There is a need for effective and well-tolerated treatments for panic disorder. If found to be effective, hydroxyzine could provide a new option for patients with this condition, potentially improving their quality of life and functioning. The results of this pilot study will inform the design of future studies and contribute to the development of evidence-based treatments for panic disorder.

ELIGIBILITY:
Inclusion Criteria:

* The study will recruit adult patients (18 years and older)
* Confirmed diagnosis of the panic disorder according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-5).
* Participants will be included if they have had at least one panic attack per week for the last four weeks,
* Have not received any pharmacological treatment for panic disorder in the past four weeks,
* Willing to discontinue any current benzodiazepine or SSRI treatment for the duration of the study.

Exclusion criteria:

* Current substance abuse or dependence,
* Medical diseases
* Psychiatric comorbidities,
* Pregnancy or lactation.

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-12-30 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Panic Disorder Severity Scale (PDSS) Mean Score | 8 weeks
  The primary outcome measure will be the change in panic disorder severity as measured by the PDSS, which will be completed at baseline, week 4, and week 8.
  The Panic Disorder Severity Scale (PDSS) is a self report scale that measures the severity of panic attacks and panic disorder symptoms. It is appropriate for use with adolescents (13+) and adults.
  The scale is a useful way of assessing overall panic disorder severity at baseline, and it provides a profile of severity of the different panic disorder symptoms. It is a good monitoring tool because it is brief and sensitive to change, and can be used to track symptoms over time.
  The scale consists of seven items, each rated on a 5-point scale. The items assess panic frequency, distress during panic, panic-focused anticipatory anxiety, phobic avoidance of situations, phobic avoidance of physical sensations, impairment in work functioning, and impairment in social functioning.

SECONDARY OUTCOMES:
Change in Clinical Global Impression Scale (CGI) Mean Score | 8 weeks
  The secondary outcome measure will be the change in clinical global impression as measured by the CGI, which will be completed at baseline, week 4, and week 8

IPD SHARING:
Plan to Share IPD: Yes